CLINICAL TRIAL: NCT03450863
Title: Impact of Fiasp® on Glycaemic Control in a Real World Population With Type 1 Diabetes Mellitus Using Flash Glucose Monitoring
Brief Title: Study on How Fiasp® Can Influence Blood Sugar Levels of type1 Diabetic Patients in Their Daily Lives, With the Help of the Freestyle Libre® Device
Acronym: GoBolus
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1218-4412; U1111-1204-0620 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fast-acting insulin aspart: Participants will receive fast-acting insulin aspart at the treating physician's discretion as part of the usual clinical practice. The prescription and use of fast-acting insulin aspart is completely independent of this study. Total study duration for the individual patient will be approximately 24 weeks.
  Interventions: Drug: Fast-acting insulin aspart

INTERVENTIONS:
Drug: Fast-acting insulin aspart — Patients will be treated with commercially available fast-acting insulin aspart as bolus insulin (multiple daily injection [MDI]) or as insulin used in the insulin pumps (continuous subcutaneous insulin infusion [CSII]). Dosing of fast-acting insulin aspart is individual and determined by the treating physician in accordance with the needs of the patient.
  Other Names: Fiasp®

SUMMARY:
The purpose of this study is to collect information about Fiasp® to evaluate how effective Fiasp® is in treating elevated blood sugar in patients with type 1 diabetes, compared with the participant's previous insulin treatment. The study will also assess how satisfied the participants are with the treatment with Fiasp® and the impact of the treatment on quality of life. The study has also been set up to learn more about how effective Fiasp® is in controlling the glucose levels during the day and night. The duration of the study is expected to be approximately 2 years. The participation is expected to be approximately 6-8 months for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedures related to recording of data according to protocol)
* The decision to initiate treatment with commercially available Fiasp® has been made by the patient and the treating physician before and independently from the decision to include the patient in this study
* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* Diagnosed with T1DM at least 1 year prior to inclusion in the study
* Stable treatment by MDI/CSII for at least 6 months prior to inclusion in the study. Stable treatment is defined as not changing the treatment method, with dose adjustments allowed
* Regular (defined as usage on a monthly basis) user of Freestyle Libre® flash glucose monitoring for at least 6 months as the only continuous glucose monitoring (CGM) system actively used and availability of a full 2 weeks sensor download as "csv" file with 80% completeness of the data (if more sensor data are available, the 2 week data closest to baseline visit will be used)
* Latest HbA1c value measured in the 3 months prior to inclusion in the study between 7.5-9.5%

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Anti-diabetic treatment intensification during the last 3 months prior to inclusion in the study. Treatment intensification is defined as adding new anti-diabetic medication to previous treatment regimen
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods. Only highly effective methods of birth control are accepted (i.e. one that results in less than 1% per year failure rate when used consistently and correctly such as implants, injectables, combined oral contraceptives, certain intrauterine devices), or sexual abstinence or a vasectomised partner

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with type 1 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
Change in Glycated Haemoglobin (HbA1c) | Baseline (week 0), end of study (week 24 ± 4 weeks after baseline)
  Measure in % point

SECONDARY OUTCOMES:
Change in Patient Reported Outcome: Impact of treatment measured by the overall score obtained from the Treatment Related Impact Measure For Diabetes (TRIM-D) questionnaire | Baseline (week 0), end of study (week 24 ± 4 weeks)
  The TRIM-D Device is an eight item measure with two domains assessing Device Bother and Device Function. This captures information on the ease of use, convenience, and handling of the device(s) used to take diabetes medication. The measure has acceptable reliability, validity and ability to detect change.
Change in Patient Reported Outcomes: Treatment satisfaction measured by the overall score obtained from the Diabetes Treatment Satisfaction Questionnaire (DTSQ) | Baseline (week 0), end of study (week 24 ± 4 weeks)
  The DTSQs questionnaire will be used to assess subject's treatment satisfaction. This instrument contains 8 items and measures the treatment for your diabetes (including insulin, tablets and/or diet) in terms of convenience, flexibility and general feelings regarding treatment.
Change in fasting plasma glucose (FPG) | Baseline (week 0), week 12 (±4 weeks)
  Measured in mmol/L
Change in fasting plasma glucose (FPG) | Baseline (week 0), end of study (week 24 ±4 weeks)
  Measured in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Schweinfurt, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/sharing-results

REFERENCES:
- [Derived] Danne T, Axel Schweitzer M, Keuthage W, Kipper S, Kretzschmar Y, Simon J, Wiedenmann T, Ziegler R. Impact of Fast-Acting Insulin Aspart on Glycemic Control in Patients with Type 1 Diabetes Using Intermittent-Scanning Continuous Glucose Monitoring Within a Real-World Setting: The GoBolus Study. Diabetes Technol Ther. 2021 Mar;23(3):203-212. doi: 10.1089/dia.2020.0360. Epub 2020 Oct 21. PMID 32924568